CLINICAL TRIAL: NCT04368117
Title: STAT: Standard Therapy Plus Active Therapy to Improve Mobility, Long-Term Activity, and Quality of Life for Severely Burn Injured Patients After Skin Graft Surgery
Brief Title: STAT: Standard Therapy Plus Active Therapy
Acronym: STAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American Burn Association (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1552346; W81XWH-19-2-0043 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2020-04-08; First posted 2020-04-29 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Burn Injury; Physical Injury; Thermal Burn
Keywords: Physical impairment
MeSH Terms: conditions — Burns | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Severely burn injured with a 15% TBSA of burn injury or larger who require a skin graft surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Therapy (ST) (Active Comparator): Patients randomized to the ST group will receive standard of care, routine burn physical therapy.
  Interventions: Behavioral: Physical Therapy
- Active Therapy (STAT) (Experimental): Patients randomized to the STAT group will receive an intensive, quantifiable, activity-based physical therapy prescription emphasizing four of the most active components of therapy: mobilization, strength training, aerobic training and functional training.
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Behavioral: Physical Therapy — Directed and prescribe physical therapy program for severely burned patients

SUMMARY:
The objective of the study is to assess the efficacy of STAT, an activity-based therapy protocol compared to standard therapy (ST) to improve functional outcome and reduce disability in patients recovering from burn injury. This randomized multi-center trial is designed with two parallel treatment groups: STAT and ST. Efficacy of the STAT protocol will be determined through comparison to the ST only group. It will be conducted at seven burn centers.

DETAILED DESCRIPTION:
This investigation is a multicenter trial involving severely burned patients. The design will be a 1:1 randomized control study comparing the rehabilitation intervention described below to current standard care in severely burned patients. This study will take place in multiple U.S. burn centers and involve adult (18 years and older) burn patient with ≥15% total body surface area (TBSA) burn who will undergo a skin graft procedure. The local burn surgeon will direct all medical and surgical treatment. The treating physician will make all clinical decisions regarding the patient.

Study Groups

Standard therapy (ST) group

Patients in the ST group will receive routine burn therapy care with no specific prescription of activities or frequency/duration of therapy. Burn therapy will begin when the patient has been medically cleared by the treating physician to begin burn therapy and when the patient undergoes surgery, therapy will halt and resume as is typical for the participating site. All burn therapy procedures will be according to what is customary and typical for the burn center. Standard therapy practices will be documented with a pre-study interview with clinicians at each participating site. Standard burn therapy typically includes interventions such as range of motion, positioning, splinting, exercise, mobilization and pressure therapy. The amount of time and types of ST interventions will be documented at the end of each session daily. Any missed or interrupted treatment time will also be documented. Post discharge home program will include what would normally be included at discharge.

Active therapy (STAT) intervention group

Patients randomized to receive STAT therapy will receive an intensive, quantifiable, activity-based protocol emphasizing four of the most active components of therapy: mobilization, strength training, aerobic training and functional training. The STAT protocol guidelines are described below. As with the ST group, STAT therapy will begin when the patient has been medically cleared by the treating physician to begin burn therapy. STAT will not be provided for any given therapy session that the patient demonstrates any of the contraindicated safety parameters defined in Table 2. When the patient undergoes surgery, the STAT protocol will be held for the day of surgery and will resume post-operative day #1 whenever possible. The STAT protocol will be implemented 30-45 minutes per day, 5 days/ per week when possible throughout the patient's care from admission until the patient is discharged from acute care with a target treatment minimum of 150 minutes per week. Over the course of a week, all four activities in the STAT protocol should be implemented when possible. Multiple activities can be addressed within one session or single activities over multiple days.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years old
2. Total TBSA of 15% or greater with at least 10% TBSA of third-degree burn
3. Potential need for a skin graft procedure determined by the local burn surgeon
4. Survivable burn injury determined by the admitting local burn surgeon on admission

Exclusion Criteria:

1. Non-survivable burn injury determined by the admitting local burn surgeon on admission
2. History of chronic renal failure requiring dialysis prior to injury
3. History of developmental delay or congenital cognitive disorders
4. Prior history of connective tissue disorders or autoimmune disease
5. Anoxic or traumatic brain injury
6. Prior history of cerebrovascular accident with residual mobility impairment
7. Neurologic injury or disease-causing mobility impairment
8. Prior history of leg amputation
9. Non-viable leg requiring amputation on admission
10. Anticipated inability to return for follow up testing after discharge
11. History of a New York Heart Association (NYHA) class IV congestive heart failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Functional exercise capacity | 3 years
  Functional exercise capacity will be determined using the 6-minute walk test (6MWT). Aerobic capacity is the primary outcome measure of this study because it evaluates the global and integrated responses of all of the systems involved in exercise (pulmonary, cardiovascular, circulatory, neuromuscular). The score of the test is the distance a patient walks in 6 minutes. Longer distance is associated with a better outcome.

SECONDARY OUTCOMES:
Long-term physical activity-functional task upper extremities | 3.5 years
  The Quick-Disabilities Assessment of the Shoulder and Hand (QuickDASH) is a questionnaire consisting of an 11-item disability/symptom scale to measure upper limb function. Score ranges from 0 (no disability) to 100 (most severe disability), so lower score associated with better outcome.
Long-term physical activity- functional task lower extremities | 3.5 years
  Lower limb function rated on a 5 point performance scale using the Higher Mobility Assessment Tool (HiMAT) Score range is from 0 to 54, with the higher score indicating better outcome.
Long-term physical activity- daily steps | 3.5 years
  Total daily steps taken will be measured using a wearable monitor in both STAT and ST
Long-term physical activity- daily distance walked | 3.5 years
  Daily distance walked will be measured using a wearable monitor in both STAT and ST
Long-term physical activity- calories used | 3.5 years
  Daily calories used will be measured using a wearable monitor in both STAT and ST
Long-term physical activity-gait quality- speed of walking | 3.5 years
  Gait parameters such as speed will be measured using the GAITrite® Platinum Plus System 14' with Logitech® Camera
Long-term physical activity-gait quality- cadence of steps | 3.5 years
  Gait parameters such as cadence will be measured using the GAITrite® Platinum Plus System 14' with Logitech® Camera
Long-term physical activity-gait quality-length of stride when walking | 3.5 years
  Gait parameters such as stride length will be measured using the GAITrite® Platinum Plus System 14' with Logitech® Camera

OTHER OUTCOMES:
Time from hospital discharge to Return to Work status | 3.5 years
  Data will be collected for both the STAT and ST group regarding number of days from hospital discharge to returning to work
Time from hospital discharge to Return to Active Duty | 3.5 years
  Data will be collected for both the STAT and ST group regarding number of days from hospital discharge to return to active duty status after burn injury.
Quality of Life - Performance of Self Care Activities of Daily Living | 3.5 years
  Data will be collected for both the STAT and ST group regarding patient reported performance of self care daily activities after burn injury, as measured by the Canadian Occupational Performance Measure (COPM). Range of score from 1-10 with 10 indicating better outcome.
Quality of Life - Performance of Leisure Activities | 3.5 years
  Data will be collected for both the STAT and ST regarding patient reported performance of leisure activities after burn injury, as measured by the Canadian Occupational Performance Measure (COPM). Range of score from 1-10 with 10 indicating better outcome.
Quality of Life - Patient reported productivity after burn injury | 3.5 years
  Data will be collected for both the STAT and ST regarding patient reported productivity after burn injury, as measured by the Canadian Occupational Performance Measure (COPM). Range of score from 1-10 with 10 indicating better outcome.
Incidence of cardiovascular complications | 3.5 years
  The incidence of cardiovascular complications will be measured in both groups.
Total Ventilator days | 3.5 years
  The number of ventilator days will be measured in both groups.
Total number of infections | 3.5 years
  The number of infections will be measured in both groups.
Hospital length of stay | 3.5 years
  Total number of hospital days will be measured in both groups.
Quality of Life Assessment: Burn Specific Health Scale (BSHS) | 3.5 years
  Burn Specific Health Scale (BSHS): The BSHS is a self-reported assessment of overall quality of life. It incorporates four overall areas that are specific for burn patients: affect and relationships, physical function, skin involvement, and work. ) Consists of 40 questions, each with score ranging from 0-4 and higher scores are associated with better outcomes.
Incidence of post surgical complications | 3.5 years
  The incidence of patients requiring repeat-skin graft procedures will be compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Soman Sen, MD, Principal Investigator — UC Davis
Locations (7):
- United States (7):
  - ValleyWise Health, Phoenix, Arizona
  - University of California Davis Medical Center-Regional Burn Center, Sacramento, California
  - Loyola University Medical Center, Maywood, Illinois
  - Health and Hospital Corporation dba Eskenazi Health, Indianapolis, Indiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - United States Army Institute of Surgical Research, Fort Sam Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available to researchers through the Burn Science Advisory Panel of the American Burn Association
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be come available 1 year after completion of study analysis and publication of initial study findings
Access Criteria: Clinical researcher with approval of use from the Burn Science Advisory Panel of the American Burn Association

REFERENCES:
- [Background] Bloomfield SA. Changes in musculoskeletal structure and function with prolonged bed rest. Med Sci Sports Exerc. 1997 Feb;29(2):197-206. doi: 10.1097/00005768-199702000-00006. PMID 9044223
- [Background] Kortebein P, Ferrando A, Lombeida J, Wolfe R, Evans WJ. Effect of 10 days of bed rest on skeletal muscle in healthy older adults. JAMA. 2007 Apr 25;297(16):1772-4. doi: 10.1001/jama.297.16.1772-b. No abstract available. PMID 17456818
- [Background] Suesada MM, Martins MA, Carvalho CR. Effect of short-term hospitalization on functional capacity in patients not restricted to bed. Am J Phys Med Rehabil. 2007 Jun;86(6):455-62. doi: 10.1097/PHM.0b013e31805b7566. PMID 17515684
- [Background] Convertino V, Hung J, Goldwater D, DeBusk RF. Cardiovascular responses to exercise in middle-aged men after 10 days of bedrest. Circulation. 1982 Jan;65(1):134-40. doi: 10.1161/01.cir.65.1.134. PMID 6796287
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Background] Convertino VA. Cardiovascular consequences of bed rest: effect on maximal oxygen uptake. Med Sci Sports Exerc. 1997 Feb;29(2):191-6. doi: 10.1097/00005768-199702000-00005. PMID 9044222
- [Background] Ferrando AA, Lane HW, Stuart CA, Davis-Street J, Wolfe RR. Prolonged bed rest decreases skeletal muscle and whole body protein synthesis. Am J Physiol. 1996 Apr;270(4 Pt 1):E627-33. doi: 10.1152/ajpendo.1996.270.4.E627. PMID 8928769
- [Background] Powers SK, Wiggs MP, Duarte JA, Zergeroglu AM, Demirel HA. Mitochondrial signaling contributes to disuse muscle atrophy. Am J Physiol Endocrinol Metab. 2012 Jul 1;303(1):E31-9. doi: 10.1152/ajpendo.00609.2011. Epub 2012 Mar 6. PMID 22395111
- [Background] Hart DW, Wolf SE, Mlcak R, Chinkes DL, Ramzy PI, Obeng MK, Ferrando AA, Wolfe RR, Herndon DN. Persistence of muscle catabolism after severe burn. Surgery. 2000 Aug;128(2):312-9. doi: 10.1067/msy.2000.108059. PMID 10923010
- [Background] Klein GL, Herndon DN, Goodman WG, Langman CB, Phillips WA, Dickson IR, Eastell R, Naylor KE, Maloney NA, Desai M, et al. Histomorphometric and biochemical characterization of bone following acute severe burns in children. Bone. 1995 Nov;17(5):455-60. doi: 10.1016/8756-3282(95)00279-1. PMID 8579956
- [Background] Klein GL, Herndon DN, Rutan TC, Sherrard DJ, Coburn JW, Langman CB, Thomas ML, Haddad JG Jr, Cooper CW, Miller NL, et al. Bone disease in burn patients. J Bone Miner Res. 1993 Mar;8(3):337-45. doi: 10.1002/jbmr.5650080311. PMID 8456588
- [Background] Kress JP. Clinical trials of early mobilization of critically ill patients. Crit Care Med. 2009 Oct;37(10 Suppl):S442-7. doi: 10.1097/CCM.0b013e3181b6f9c0. PMID 20046133
- [Background] Burtin C, Clerckx B, Robbeets C, Ferdinande P, Langer D, Troosters T, Hermans G, Decramer M, Gosselink R. Early exercise in critically ill patients enhances short-term functional recovery. Crit Care Med. 2009 Sep;37(9):2499-505. doi: 10.1097/CCM.0b013e3181a38937. PMID 19623052
- [Background] Kayambu G, Boots R, Paratz J. Early physical rehabilitation in intensive care patients with sepsis syndromes: a pilot randomised controlled trial. Intensive Care Med. 2015 May;41(5):865-74. doi: 10.1007/s00134-015-3763-8. Epub 2015 Apr 8. PMID 25851383
- [Background] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Bailey P, Thomsen GE, Spuhler VJ, Blair R, Jewkes J, Bezdjian L, Veale K, Rodriquez L, Hopkins RO. Early activity is feasible and safe in respiratory failure patients. Crit Care Med. 2007 Jan;35(1):139-45. doi: 10.1097/01.CCM.0000251130.69568.87. PMID 17133183
- [Background] Stiller K. Physiotherapy in intensive care: an updated systematic review. Chest. 2013 Sep;144(3):825-847. doi: 10.1378/chest.12-2930. PMID 23722822
- [Background] Nydahl P, Sricharoenchai T, Chandra S, Kundt FS, Huang M, Fischill M, Needham DM. Safety of Patient Mobilization and Rehabilitation in the Intensive Care Unit. Systematic Review with Meta-Analysis. Ann Am Thorac Soc. 2017 May;14(5):766-777. doi: 10.1513/AnnalsATS.201611-843SR. PMID 28231030
- [Background] Lorello DJ, Peck M, Albrecht M, Richey KJ, Pressman MA. Results of a prospective randomized controlled trial of early ambulation for patients with lower extremity autografts. J Burn Care Res. 2014 Sep-Oct;35(5):431-6. doi: 10.1097/BCR.0000000000000014. PMID 25100538
- [Background] Nedelec B, Serghiou MA, Niszczak J, McMahon M, Healey T. Practice guidelines for early ambulation of burn survivors after lower extremity grafts. J Burn Care Res. 2012 May-Jun;33(3):319-29. doi: 10.1097/BCR.0b013e31823359d9. PMID 21959211
- [Background] Parry I, Forbes L, Lorello D, Benavides L, Calvert C, Hsu SC, Chouinard A, Godleski M, Helm P, Holavanahalli RK, Kemp-Offenberg J, Ruiz CE, Shon R, Schneider JC, Shetler M, Suman OE, Nedelec B. Burn Rehabilitation Therapists Competency Tool-Version 2: An Expansion to Include Long-Term Rehabilitation and Outpatient Care. J Burn Care Res. 2017 Jan/Feb;38(1):e261-e268. doi: 10.1097/BCR.0000000000000364. PMID 27359189
- [Background] Richard R, Santos-Lozada AR. Burn Patient Acuity Demographics, Scar Contractures, and Rehabilitation Treatment Time Related to Patient Outcomes: The ACT Study. J Burn Care Res. 2017 Jul/Aug;38(4):230-242. doi: 10.1097/BCR.0000000000000490. PMID 28644206
- [Background] Deng H, Chen J, Li F, Li-Tsang CW, Liu Q, Ma X, Ao M, Chen N, Zhou Y, Zhong X, Chen Z, Cao L, He G, Wu J. Effects of mobility training on severe burn patients in the BICU: A retrospective cohort study. Burns. 2016 Nov;42(7):1404-1412. doi: 10.1016/j.burns.2016.07.029. Epub 2016 Aug 29. PMID 27595451
- [Background] Wells NJ, Boyle JC, Snelling CF, Carr NJ, Courtemanche DJ. Lower extremity burns and Unna paste: can we decrease health care costs without compromising patient care? Can J Surg. 1995 Dec;38(6):533-6. PMID 7497369
- [Background] Parry I, Painting L, Bagley A, Kawada J, Molitor F, Sen S, Greenhalgh DG, Palmieri TL. A Pilot Prospective Randomized Control Trial Comparing Exercises Using Videogame Therapy to Standard Physical Therapy: 6 Months Follow-Up. J Burn Care Res. 2015 Sep-Oct;36(5):534-44. doi: 10.1097/BCR.0000000000000165. PMID 26335108
- [Background] Parry IS, Bagley A, Kawada J, Sen S, Greenhalgh DG, Palmieri TL. Commercially available interactive video games in burn rehabilitation: therapeutic potential. Burns. 2012 Jun;38(4):493-500. doi: 10.1016/j.burns.2012.02.010. Epub 2012 Mar 3. PMID 22385641
- [Background] Parry I, Carbullido C, Kawada J, Bagley A, Sen S, Greenhalgh D, Palmieri T. Keeping up with video game technology: objective analysis of Xbox Kinect and PlayStation 3 Move for use in burn rehabilitation. Burns. 2014 Aug;40(5):852-9. doi: 10.1016/j.burns.2013.11.005. Epub 2013 Dec 2. PMID 24296065
- [Background] Richard RL, Hedman TL, Quick CD, Barillo DJ, Cancio LC, Renz EM, Chapman TT, Dewey WS, Dougherty ME, Esselman PC, Forbes-Duchart L, Franzen BJ, Hunter H, Kowalske K, Moore ML, Nakamura DY, Nedelec B, Niszczak J, Parry I, Serghiou M, Ward RS, Holcomb JB, Wolf SE. A clarion to recommit and reaffirm burn rehabilitation. J Burn Care Res. 2008 May-Jun;29(3):425-32. doi: 10.1097/BCR.0b013e318171081d. PMID 18388581
- [Background] Grisbrook TL, Stearne SM, Reid SL, Wood FM, Rea SM, Elliott CM. Demonstration of the use of the ICF framework in detailing complex functional deficits after major burn. Burns. 2012 Feb;38(1):32-43. doi: 10.1016/j.burns.2011.04.001. Epub 2011 Nov 12. PMID 22079536
- [Background] Cucuzzo NA, Ferrando A, Herndon DN. The effects of exercise programming vs traditional outpatient therapy in the rehabilitation of severely burned children. J Burn Care Rehabil. 2001 May-Jun;22(3):214-20. doi: 10.1097/00004630-200105000-00006. PMID 11403243
- [Background] Bohannon RW, Crouch R. Minimal clinically important difference for change in 6-minute walk test distance of adults with pathology: a systematic review. J Eval Clin Pract. 2017 Apr;23(2):377-381. doi: 10.1111/jep.12629. Epub 2016 Sep 4. PMID 27592691
- [Background] Oostdam N, van Poppel MN, Eekhoff EM, Wouters MG, van Mechelen W. Design of FitFor2 study: the effects of an exercise program on insulin sensitivity and plasma glucose levels in pregnant women at high risk for gestational diabetes. BMC Pregnancy Childbirth. 2009 Jan 5;9:1. doi: 10.1186/1471-2393-9-1. PMID 19123930
- [Background] Jarrett M, McMahon M, Stiller K. Physical outcomes of patients with burn injuries--a 12 month follow-up. J Burn Care Res. 2008 Nov-Dec;29(6):975-84. doi: 10.1097/BCR.0b013e31818ba172. PMID 18849834
- [Background] Willis CE, Grisbrook TL, Elliott CM, Wood FM, Wallman KE, Reid SL. Pulmonary function, exercise capacity and physical activity participation in adults following burn. Burns. 2011 Dec;37(8):1326-33. doi: 10.1016/j.burns.2011.03.016. Epub 2011 May 6. PMID 21530086
- [Background] Ganio MS, Pearson J, Schlader ZJ, Brothers RM, Lucas RA, Rivas E, Kowalske KJ, Crandall CG. Aerobic Fitness Is Disproportionately Low in Adult Burn Survivors Years After Injury. J Burn Care Res. 2015 Jul-Aug;36(4):513-9. doi: 10.1097/BCR.0b013e3182a22915. PMID 24043241
- [Background] Mathie MJ, Coster AC, Lovell NH, Celler BG. Accelerometry: providing an integrated, practical method for long-term, ambulatory monitoring of human movement. Physiol Meas. 2004 Apr;25(2):R1-20. doi: 10.1088/0967-3334/25/2/r01. PMID 15132305
- [Background] Grisbrook TL, Reid SL, Elliott CM, Elliott BC, Edgar DW, Wood FM. Lower limb functional outcome assessment following burn injury: a novel use for 3D laboratory-based movement analysis. Burns. 2010 May;36(3):e24-30. doi: 10.1016/j.burns.2009.01.006. Epub 2009 May 12. No abstract available. PMID 19442449
- [Background] Gummesson C, Ward MM, Atroshi I. The shortened disabilities of the arm, shoulder and hand questionnaire (QuickDASH): validity and reliability based on responses within the full-length DASH. BMC Musculoskelet Disord. 2006 May 18;7:44. doi: 10.1186/1471-2474-7-44. PMID 16709254
- [Background] Finlay V, Phillips M, Wood F, Hendrie D, Allison GT, Edgar D. Enhancing the clinical utility of the burn specific health scale-brief: not just for major burns. Burns. 2014 Mar;40(2):328-36. doi: 10.1016/j.burns.2013.07.005. Epub 2013 Sep 14. PMID 24045070
- [Background] Tyack Z, Ziviani J, Kimble R, Plaza A, Jones A, Cuttle L, Simons M. Measuring the impact of burn scarring on health-related quality of life: Development and preliminary content validation of the Brisbane Burn Scar Impact Profile (BBSIP) for children and adults. Burns. 2015 Nov;41(7):1405-19. doi: 10.1016/j.burns.2015.05.021. Epub 2015 Oct 1. PMID 26421693
- [Background] Clark DE, Lowman JD, Griffin RL, Matthews HM, Reiff DA. Effectiveness of an early mobilization protocol in a trauma and burns intensive care unit: a retrospective cohort study. Phys Ther. 2013 Feb;93(2):186-96. doi: 10.2522/ptj.20110417. Epub 2012 Aug 9. PMID 22879442
- [Background] Kmetic A, Joseph L, Berger C, Tenenhouse A. Multiple imputation to account for missing data in a survey: estimating the prevalence of osteoporosis. Epidemiology. 2002 Jul;13(4):437-44. doi: 10.1097/00001648-200207000-00012. PMID 12094099
- [Background] Resseguier N, Giorgi R, Paoletti X. Sensitivity analysis when data are missing not-at-random. Epidemiology. 2011 Mar;22(2):282. doi: 10.1097/EDE.0b013e318209dec7. No abstract available. PMID 21293212